CLINICAL TRIAL: NCT04776122
Title: Breathing and CBT Platform Usability Take-home Study
Brief Title: Usability of a Breathing-CBT Platform (CBT = Cognitive Behavioural Therapy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: eLB0409-316
Record Dates: First submitted 2020-04-06; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Breathing, Mouth
MeSH Terms: conditions — Mouth Breathing | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control with no device (Active Comparator): Breathing performed with no device
  Interventions: Other: No device
- Therapy - device assisted breathing (Experimental): Breathing performed with device
  Interventions: Device: Therapy

INTERVENTIONS:
Device: Therapy — Device-assisted breathing for relaxation
  Arms: Therapy - device assisted breathing
Other: No device — Breathing platform without device
  Arms: Control with no device

SUMMARY:
The study will examine the usability of a breathing platform in the home environment. It will be a randomized, open-label crossover study of 10 participants who will complete the CBT and breathing components in their home, prior to sleeping. Usability will be measured by scores assigned by participants. Qualitative feedback and compliance information will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing to give written, informed consent
* Participants are healthy adults
* Participants are able to comprehend and speak English
* Participants are at least 18 years of age

Exclusion Criteria:

* Participants who are/may be pregnant or lactating
* Participant that have a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury)
* Participants who are unsuitable for the inclusion at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Ease of use | 8 days
  Participants will complete a questionnaire rating how easy it was to use and sleep with the device providing assistance to their breathing patterns

SECONDARY OUTCOMES:
Compliance | 8 days
  Frequency of use, as assessed by a short questionnaire asking how often patients used the device

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Armitstead, Principal Investigator — ResMed
Locations (1):
- ResMed Ltd, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No